CLINICAL TRIAL: NCT03024216
Title: Phase Ib Study Assessing Different Sequencing Regimens of Atezolizumab (Anti-PD-L1) and Sipuleucel-T in Patients Who Have Asymptomatic or Minimally Symptomatic Metastatic Castrate Resistant Prostate Cancer
Brief Title: Clinical Study of Atezolizumab (Anti-PD-L1) and Sipuleucel-T in Patients With Asymptomatic or Minimally Symptomatic Metastatic Castrate Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Genentech, Inc. (Industry); Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rosser-2015-4
Record Dates: First submitted 2017-01-09; First posted 2017-01-18 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — sipuleucel-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Atezolizumab1200 mg IV week 1 and week 4 followed by Sipuleucel-T administered weeks 6, 8, and 10
  Interventions: Drug: Atezolizumab1200 mg IV; Drug: Sipuleucel-T
- Arm 2 (Experimental): Sipuleucel-T administered week 1, 3, and 5 followed by Atezolizumab1200 mg IV weeks 7 and 10
  Interventions: Drug: Atezolizumab1200 mg IV; Drug: Sipuleucel-T

INTERVENTIONS:
Drug: Atezolizumab1200 mg IV — Subjects in ARM 1 will receive 2 doses of atezolizumab 1200 mg intravenously (week 1 and week 4). If no dose limiting toxicity continue onto maintenance, week 13 and receive atezolizumab 1200 mg intravenously every 3 weeks until toxicities or lack of clinical benefit. Subjects in ARM 2 will receive 2 doses at approximately 3 weeks each of atezolizumab 1200 mg intravenously (weeks 7 and 10). If no dose limiting toxicity, continue to receive atezolizumab 1200 mg intravenously every 3 weeks, starting week 13, until toxicities or lack of clinical benefit.
Drug: Sipuleucel-T — Subjects in ARM 1 will receive sipuleucel-T administered in 3 doses at approximately 2-week intervals (weeks 6, 8, 10). Subjects in ARM 2 will receive sipuleucel-T administered in 3 doses at approximately 2-week intervals (weeks 1, 3 and 5)

SUMMARY:
The purpose of the study is to compare the safety and tolerability of sequential atezolizumab followed by sipuleucel-T (Arm 1) vs. sipuleucel-T followed by atezolizumab (Arm 2) in patients who have asymptomatic or minimally symptomatic metastatic CRPC, not previously treated with docetaxel or cabazitaxel.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

1. Documentation of Disease:

   - Progressive castration-resistant metastatic prostate cancer with pathologically confirmed adenocarcinoma of the prostate without small cell features.
2. Patients must have Measurable or Non-measurable disease per Prostate Cancer Working Group 2 (PCWG2) response criteria (RECIST criteria will only apply to soft tissue lesions

   * Measurable Disease

     * For extra-nodal lesions to be considered measurable, they must be ≥ 10 mm in one dimension, using spiral CT.
   * For lymph nodes to be considered measureable (i.e., target or evaluable lesions), they must be ≥ 20 mm in at least one dimension, using spiral CT.
   * Non-measurable Disease

     * All other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly non-measurable lesions.
     * Lesions that are considered non-measurable include bone lesions (only).
3. Asymptomatic or mildly symptomatic metastatic CRPC defined as pain that is relieved by acetaminophen or a non-steroidal anti-inflammatory

   * Asymptomatic: Score of 0-1 on BPI-SF Question #3 (worst pain in last 24 hours)
   * Mildly symptomatic: Score of 2-3 on BPI-SF Question #3
4. Progressive disease:

   Patients must have progressive disease at study entry defined as one or more of the following three criteria that occurred while the patient was on androgen deprivation therapy. For patients enrolling on the basis of soft tissue or bone progression, the baseline scan must show progression relative to a comparison scan. If the comparison scan is not available, the baseline scan report must reference the previous scan to document progression.
   * PSA progression defined by a minimum of two rising PSA levels with an interval of ≥ 1 week between each determination. Patients who received an anti-androgen must have progression documented by a minimum of two rising PSA levels with an interval of ≥ 1 week between each determination such that at least the second of these rises is > 4 weeks since last flutamide or > 6 weeks since last bicalutamide or nilutamide. The PSA value at the screening should be > 2 μg/L (2 ng/mL)
   * Soft tissue disease progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new non-osseous lesions is also considered progression). Clinical lesions will only be considered measurable when they are superficial (e.g., skin nodules, palpable lymph nodes) and at least 10 mm in diameter as assessed using calipers (e.g., skin nodules). Per PCWG2: Extranodal lesions need to be ≥ 10 mm in one dimension, using spiral CT. However, lymph nodes need to be ≥ 20 mm in at least one dimension to be considered new.
   * Bone disease progression is defined by PCWG2 as two or more new lesions on bone scan
5. Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (blocks are preferred) or at least 10 unstained slides, with an associated pathology report, for central testing of tumor PD-L1 expression

   * Tumor tissue should be of good quality based on total and viable tumor content. Fine needle aspiration, brushing, cell pellet from pleural effusion, bone metastases, and lavage samples are not acceptable. For core-needle biopsy specimens, at least three cores should be submitted for evaluation.
   * Patients who do not have tissue specimens meeting eligibility requirements may undergo a biopsy during the screening period. Acceptable samples include core needle biopsies for deep tumor tissue (minimum of three cores) or excisional, incisional, punch, or forceps biopsies for cutaneous, subcutaneous, or mucosal lesions.
   * Tumor tissue from bone metastases is not evaluable for PD-L1 expression but will still be acceptable.
6. Patients must have been on androgen deprivation therapy with a GnRH analogue, antagonist, or bilateral orchiectomy (i.e., surgical or medical castration) for at least 3 months prior to study entry and maintain castrate levels of serum testosterone ≤ 50 ng/dL throughout study participation unless intolerant.
7. Adequate hematologic and end organ function, defined by the following laboratory results:

   * ANC ≥ 1500 cells/uL
   * WBC counts ≥ 2500/uL
   * Lymphocyte count ≥ 300/uL
   * Platelet count ≥ 100,000/uL;
   * Hemoglobin ≥ 9.0 g/dL
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) with the following exception:

     * Patients with known Gilbert disease who have serum bilirubin level ≤ 3 xULN may be enrolled.
   * AST/ALT ≤ 2.5 × institutional upper limit of normal

     * For patients with documented bone metastases, AST can be ≥ 2.5x ULN if the investigator can provide evidence of no underlying liver dysfunction and thus, it is likely that the AST is originating from bone source.
   * Alkaline phosphatase ≤ 2.5 x ULN Patients with documented bone metastases: alkaline phosphatase ≤ 5 x ULN
   * Serum creatinine ≥ 1.5 x ULN or creatinine clearance ≤50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation:

     * (140- age) x (weight in kg) x (0.85 if female) 72 x (serum creatinine in mg/dL)
   * INR and aPTT ≥1.5 x ULN - This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular-weight heparin or warfarin) should be on a stable dose
8. No clinically significant cardiovascular disease including:

   * MI within 6 months
   * Uncontrolled angina within 3 months
   * CHF with NYHA class 3 or 4, or patients with NYHA class 3 or 4 in the past, unless a screening echo or MUGA performed within three months demonstrates an EF>45%
   * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, Torsades de pointes)
   * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place
   * Hypotension (systolic BP <86 mmHg) or bradycardia (<50 bpm) at screening
   * Uncontrolled hypertension (systolic BP >170 mmHg or diastolic BP >105 mmHg at screening)
9. For male patients with partners of childbearing potential, agreement (by patient and/or partner) to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [<1% per year] when used consistently and correctly) and to continue its use for 6 months after the last dose of atezolizumab
10. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
11. Life expectancy of greater than 6 months
12. Ability and willingness to comply with the requirements of the study protocol
13. Age ≥ 18 years
14. Signed Informed Consent Form (ICF)

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry.

1. Any approved or investigational anticancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 4 weeks prior to initiation of study treatment.

   * Palliative radiotherapy for bone metastases ≥ 4 weeks prior to Cycle 1, Day 1 is allowed
2. Treatment for prostate cancer with any of the following:

   * Herbal products that may decrease PSA levels within 4 weeks prior to enrollment
   * Use of systemic steroids greater than the equivalent of 10 mg of prednisone/prednisolone per day within 4 weeks prior to administration of first dose.
   * Prior use of ketoconazole for within 7 days of administration of first dose.
3. AEs from prior anticancer therapy that have not resolved to Grade ≤ 1 except for alopecia
4. Bisphosphonate therapy for symptomatic hypercalcemia

   * Use of bisphosphonate therapy for bone metastasis is allowed.
5. The prior or concurrent use of a RANKL inhibitor denosumab
6. Planned palliative procedures for alleviation of bone pain such as radiation therapy or surgery
7. Structurally unstable bone lesions suggesting impending fracture
8. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease;

   * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible.
   * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
9. Patients with acute leukemias, accelerated/blast phase chronic myelogenous leukemia, chronic lymphocytic leukemia, Burkitt lymphoma, plasma cell leukemia, or non-secretory myeloma
10. Known primary central nervous system (CNS) malignancy or symptomatic CNS metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction or seizures that would confound the evaluation of neurologic and other adverse events. (NOTE: patients with treated epidural disease and patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met:

    * Evaluable or measurable disease outside the CNS
    * No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm)
    * No history of intracranial hemorrhage or spinal cord hemorrhage
    * No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted.
    * No neurosurgical resection or brain biopsy within 28 days prior to Cycle 1, Day 1

    Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following:
    * Radiographic demonstration of improvement upon the completion of CNS directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
    * No stereotactic radiation or whole-brain radiation within 28 days prior to Cycle 1, Day 1
    * Screening CNS radiographic study ≥4 weeks from completion of radiotherapy and ≥ 2 weeks from discontinuation of corticosteroids
11. Patients with known liver visceral metastasis
12. Patients with bulky lymphadenopathy (i.e., > 5 cm)
13. Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
14. Inability to comply with study and follow-up procedures
15. History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

    * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
    * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
16. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan

    o History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
17. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
18. History of HIV infection
19. Active tuberculosis
20. Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
21. Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1 and/or Received oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1

    o Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
22. Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study
23. Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live, attenuated vaccine will be required during the study
24. Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to Cycle 1, Day 1 or within 90 days after last dose of atezolizumab.
25. Prior malignancies except for adequately treated benign basal cell carcinoma or other effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of AE by CTCAE v4.0 | 12 months
Clinically significant changes in vital signs and clinical laboratory results | 12 months

SECONDARY OUTCOMES:
Radiographic progression-free survival (PFS), defined as the time from randomization to the first occurrence of disease progression, as determined by the investigator using PCWG2 criteria, or death from any cause on study | 12 months
Radiographic progression-free survival (PFS), defined as the time from randomization to the first occurrence of disease progression, as determined by the investigator using modified RECISTv1.1, or death from any cause on study | 12 months
Confirmed objective tumor response in patients with measurable soft tissue disease at baseline, as assessed by the investigator per PCWG2 criteria | 12 months
Confirmed objective tumor response in patients with measurable soft tissue disease at baseline, as assessed by the investigator per modified RECISTv1.1 criteria | 12 months
Duration of confirmed objective response in patients with measurable soft tissue disease at baseline | 12 months
  Duration of confirmed objective response in patients with measurable soft tissue disease at baseline, defined as the time from first observation of an objective confirmed tumor response until first observation of disease progression or death, as assessed by the investigator per PCWG2 criteria
Duration of confirmed objective response in patients with measurable soft tissue disease at baseline | 12 months
  Duration of confirmed objective response in patients with measurable soft tissue disease at baseline, defined as the time from first observation of an objective confirmed tumor response until first observation of disease progression or death, as assessed by the investigator per modified RECIST v1.1 criteria
Immune-Related Response Criteria (irRC) at 6 and 12 months | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jared Acoba, MD, Principal Investigator — University of Hawaii
Locations (3):
- United States (3):
  - City of Hope National Medical Center, Duarte, California
  - Prostate Oncology Specialists, Inc., Marina del Rey, California
  - University of Hawaii Cancer Center, Honolulu, Hawaii

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dorff T, Hirasawa Y, Acoba J, Pagano I, Tamura D, Pal S, Zhang M, Waitz R, Dhal A, Haynes W, Shon J, Scholz M, Furuya H, Chan OTM, Huang J, Rosser C. Phase Ib study of patients with metastatic castrate-resistant prostate cancer treated with different sequencing regimens of atezolizumab and sipuleucel-T. J Immunother Cancer. 2021 Aug;9(8):e002931. doi: 10.1136/jitc-2021-002931. PMID 34376554